CLINICAL TRIAL: NCT04345783
Title: A Study on the Efficacy and Safety of Camrelizumab for Injection, Apatinib Mesylate and Tegio for First-line Refractory Patients With Advanced Gastric Cancer
Brief Title: Efficacy and Safety of Camrelizumab for Injection, Apatinib Mesylate and Tegio for First-line Refractory Patients With Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhongtao Zhang, Professor, Beijing Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BFH-CamrelizumabCombo3
Record Dates: First submitted 2020-04-12; First posted 2020-04-14 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — camrelizumab; Injections; apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab+Apatinib Mesylate+Tegio (Experimental)
  Interventions: Drug: Camrelizumab for injection, apatinib mesylate and tegio

INTERVENTIONS:
Drug: Camrelizumab for injection, apatinib mesylate and tegio — Camrelizumab for injection: fixed dose of 200 mg, ivgtt for 30 minutes, given on D1, repeat for every 3 weeks; Apatinib mesylate: 250 mg, p.o, qd; Tegio capsule: p.o., bid, D1-14, repeat for every 21 days.

SUMMARY:
This is a prospective, single-center, single-arm, open-label clinical study, aiming at evaluating the efficacy and safety of camrelizumab for injection, apatinib mesylate and tegio for first-line refractory patients with advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged 18-75;
* 2. ECOG score 0-2;
* 3. Pathologically diagnosed late-stage adenocarcinoma of stomach or gastroesophageal junction, with extra-gastric measurable lesions (spiral CT scan≥10 mm, meeting RECIST 1.1 criteria);
* 4. Patients with locally advanced or metastatic gastric or gastroesophageal junction adenocarcinoma that are refractory to first-line chemotherapy;
* 5. Patients who received no previous treatment with apatinib or other VEGFR inhibitors, e.g. sorafenib and sunitinib;
* 6. Normal blood routine examination: Neutrophil count ≥ 1.5 × 109 / L; Hemoglobin ≥ 80 g / L; Platelet count ≥ 100 × 109 / L; Total bilirubin ≤ 1.5 × ULN; ALT, AST≤2.5×ULN；
* 7. Without severe dysfunction of heart, lung, liver or kidney, without jaundice and digestive tract obstruction, and without acute infection.

Exclusion Criteria:

* 1. KPS < 60, or estimated survival < 3 months;
* 2. Patients with cardiovascular and cerebrovascular events within half a year; patients with uncontrollable hypertension (systolic pressure > 140 mmHg, diastolic pressure > 90 mmHg), coronary heart disease above grade I, arrhythmia (including QTc interval prolongation > 450 ms in men, 470 MS in women) and grade I cardiac dysfunction; patients positive of urine albumin;
* 3. Patients with definite tendency of gastrointestinal bleeding, local active ulcer focus, and occult blood in stool (+ +); patients with history of black stool and hematemesis within 2 months;
* 4. Abnormal coagulation (INR > 1.5, APTT > 1.5 ULN), with bleeding tendency;
* 5. Patients with factors that can affect the absorption of oral-intake drugs (such as inability to swallow, nausea, vomiting, chronic diarrhea and intestinal obstruction, etc.);
* 6. Patients with nervous and mental diseases or with severe infection;
* 7. Pregnant or lactating women or those who have fertility requirements during the study period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
DFS | 3 years
  disease free survival
OS | 3 years
  overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Wei Deng, M.D., Study Director — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: from 2022.12 on

REFERENCES:
- [Derived] Jing C, Wang J, Zhu M, Bai Z, Zhao B, Zhang J, Yin J, Yang X, Liu Z, Zhang Z, Deng W. Camrelizumab combined with apatinib and S-1 as second-line treatment for patients with advanced gastric or gastroesophageal junction adenocarcinoma: a phase 2, single-arm, prospective study. Cancer Immunol Immunother. 2022 Nov;71(11):2597-2608. doi: 10.1007/s00262-022-03174-9. Epub 2022 Mar 18. PMID 35304622